CLINICAL TRIAL: NCT05823194
Title: The Evaluation of Infertility and Pregnancy Outcomes, as Well as the Assessment of Quality of Life Using WHOQoL and FertiQoL, in Cases of Gynecological Malignancies That Have Undergone Fertility-sparing Surgery(FSS)
Brief Title: Infertility and Pregnancy Outcomes of Fertility Spared Gynecological Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nazli Albayrak, PGY-4 Ob/Gyn resident, MD, Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-17/10
Record Dates: First submitted 2023-03-18; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Fertility Disorders; Gynecologic Cancer
Keywords: fertility sparing; gynecologic malignancy; quality of life; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: The study included a comprehensive evaluation of the participants' medical history, surgical procedures, oncological treatment, and fertility preservation methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fertility spared gynecologic cancer diagnosed women (Other): Participants recruited from a tertiary care hospital, and women diagnosed with gynecological malignancies (e.g. cervical, ovarian, endometrial cancer) who underwent fertility-sparing surgery between 2010 and 2022.
  Interventions: Procedure: Fertility sparing surgery

INTERVENTIONS:
Procedure: Fertility sparing surgery — Sparing the uterus and/or ovaries of the patients suffering from gynecologic malignancies to keep the patients' fertility

SUMMARY:
FSS which aims to preserve a woman's fertility while still effectively treating the cancer, has become an increasingly popular option for young women diagnosed with these types of cancers. It is important to assess how FSS affects a woman's reproductive health, sexual function, psychological well-being, and overall quality of life. This research aims to provide valuable insights into the long-term effects of FSS on a woman's life, and can help healthcare providers make informed decisions about the best treatment options for their patients.

DETAILED DESCRIPTION:
This is a prospective cohort study that aims to evaluate the infertility and pregnancy outcomes, as well as the quality of life of women who underwent fertility-sparing surgery for gynecological malignancies. The study included a comprehensive evaluation of the participants' medical history, surgical procedures, oncological treatment, and fertility preservation methods. Participants recruited from a tertiary care hospital, and women diagnosed with gynecological malignancies (e.g. cervical, ovarian, endometrial cancer) who underwent fertility-sparing surgery between 2010 and 2022. Women who have undergone total hysterectomy, bilateral salpingo-oophorectomy, or adjuvant oncological treatment were excluded from the study. Participants were contacted by phone and asked to complete questionnaires to assess their quality of life using the WHOQoL-BREF and FertiQoL scales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gynecologic cancer, and being fertile in the meantime
* Applying directly to gynecologic oncology department
* Demand of preserving the fertility

Exclusion Criteria:

* Having hysterectomy prior to the diagnosis
* Having bilateral ooferectomy prior to the diagnosis
* Being in menopause
* Not accepting to fill the survey
* High stage disease which is not able to have FSS

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of pregnancy of patients received FSS | In 12 years after FSS
  Incidence and rate of patients getting pregnant after FSS
Rate of pregnancy after FSS of patients seeking fertility by applying to IVF clinics | In 12 years after FSS
  Rate of patients referring to IVF clinic after FSS

SECONDARY OUTCOMES:
Satisfaction assesed by WHO-QoL Bref and decision-regret scale after FSS | 12 years
  % of patients' satisfaction via Quality of life after the surgery, and decision-regret analysis regarding to fertility sparing by the validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: NAZLI ALBAYRAK, MD, Principal Investigator — Acibdem University
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Result] Wang A, Cui G, Jin C, Wang Y, Tian X. Multicenter research on tumor and pregnancy outcomes in patients with early-stage cervical cancer after fertility-sparing surgery. J Int Med Res. 2019 Jul;47(7):2881-2889. doi: 10.1177/0300060519845974. Epub 2019 May 22. PMID 31115262
- [Result] Gullo G, Etrusco A, Cucinella G, Perino A, Chiantera V, Lagana AS, Tomaiuolo R, Vitagliano A, Giampaolino P, Noventa M, Andrisani A, Buzzaccarini G. Fertility-Sparing Approach in Women Affected by Stage I and Low-Grade Endometrial Carcinoma: An Updated Overview. Int J Mol Sci. 2021 Oct 31;22(21):11825. doi: 10.3390/ijms222111825. PMID 34769256
- [Result] Kovacs P. Fertility preservation in reproductive age women with cancer. J Obstet Gynaecol India. 2014 Dec;64(6):381-7. doi: 10.1007/s13224-014-0626-0. Epub 2014 Oct 30. PMID 25489139
- [Result] Levine JM, Kelvin JF, Quinn GP, Gracia CR. Infertility in reproductive-age female cancer survivors. Cancer. 2015 May 15;121(10):1532-9. doi: 10.1002/cncr.29181. Epub 2015 Feb 3. PMID 25649243